CLINICAL TRIAL: NCT04400422
Title: Experience of Using Lipano in Children With LCHAD (Long Chain Fatty Acid Oxidation Disorder)
Brief Title: Experience of Using Lipano in Children With Fatty Acid Oxidation Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Schär AG / SPA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Lipano 1 - Case
Record Dates: First submitted 2020-05-18; First posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Fatty Acid Oxidation Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lipano MCT formula (Experimental): Kanso Lipano will be consumed daily for 3 months each to assess tolerability and compliance
  Interventions: Dietary Supplement: Lipano formula

INTERVENTIONS:
Dietary Supplement: Lipano formula — Subjects will be asked to take an MCT infant formula to assess the tolerability, compliance and overall acceptability of the product for patient with LCHAD

SUMMARY:
This is a market research, observational study to evaluate the tolerability and acceptability of an MCT based formula for infants and young people with long chain fatty acid oxidation disorder from birth to 18 months. Patients with a confirmed diagnosis of a fatty acid oxidation disorder, which requires a specialist diet including MCT will be included in this study

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a fatty acid oxidation disorder requiring a ketogenic or a specialist diet as part of their treatment, which includes MCT.
* Patients from birth to 18 months
* Written informed consent obtained from patient or parental caregiver

Exclusion Criteria:

* Presence of serious concurrent illness
* Investigator's uncertainty about the willingness or ability of the patient to comply with the protocol requirements
* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study.
* Any patients having taken antibiotics over the previous 2 weeks leading up to the study
* Patients over 18 months of age

Max Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal tolerance: questionnaire | 90 days
  Daily questionnaire detailing any GI symptoms, severity and change from usual The collection of daily data about the gastrointestinal tolerance of the product
Product compliance | 90 days
  Daily questionnaire on amounts offered and amounts actually consumed, compared to recommended amount.
Product palatability | 90 days
  Questionnaire data captured to evaluate taste
Product acceptability | 90 days
  Brief tick-box questionnaire on overall liking and acceptability of product

SECONDARY OUTCOMES:
Biochemistry stability - creatine kinase | 90 days
  creatine kinase will be monitored
Biochemistry stability - liver enzymes | 90 days
  liver enzymes will be monitored
Anthropometry 1 | 90 days
  weight in g monitored to check growth
Anthropometry 2 | 90 days
  height in cm monitored to check growth

CONTACTS AND LOCATIONS:
Locations (1):
- Russian Children's Hospital Center for Orphan Diseases, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
This study will be used to demonstrate acceptability for registration and reimbursement of these foods for special medical purposes.